CLINICAL TRIAL: NCT04969757
Title: Evaluation of the Use of the Predigraft Platform (a Remote Monitoring Solution for Predicting Kidney Graft Survival) in Kidney Transplant Patients
Brief Title: Use of Predigraft in Kidney Transplant Patients
Acronym: PREDIGRAFT2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP210379
Record Dates: First submitted 2021-06-17; First posted 2021-07-21 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Kidney Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Predigraft (Experimental): Patients in the interventional arm will use Predigraft (Class 1 medical device under MDD 93/42/EEC Cibiltech Society) to receive therapeutic education content (videos, facts sheets, short messages, questionnaires), exchange documents with their doctors and interact via messaging with them.
  Physicians will be able to calculate their iBox score to predict their patients' allograft survival at 3, 5 and 7 years.
  Interventions: Device: Predigraft group

INTERVENTIONS:
Device: Predigraft group — Patients in the interventional arm will use Predigraft (Class 1 medical device under MDD 93/42/EEC Cibiltech Society) to receive therapeutic education content (videos, facts sheets, short messages, questionnaires), exchange documents with their doctors and interact via messaging with them.
  Physicians will be able to calculate their iBox score to predict their patients' allograft survival at 3, 5 and 7 years.

SUMMARY:
Kidney transplantation is the treatment of choice for end-stage renal disease in terms of morbidity, mortality, and cost-benefit ratio. Graft loss is mainly related to the occurrence of rejection. Hence the importance of regular monitoring to check that the graft is functioning properly, to adapt immunosuppressive treatments and to check for side effects related to the immunosuppressed state.

In conventional management, the patient is seen at regular intervals (ranging from 2 weeks to 3 months) in the referral transplant centre with recourse to hospitalisation if necessary. In the context of the COVID-19 pandemic, in order to reduce the risks of contamination, teleconsultations have been proposed to replace face-to-face consultations. Predigraft software facilitates remote patient assessment. This software provides an estimate of the probability of renal graft survival at 3, 5 and 7 years of the assessment based on an algorithm developed and validated by the U970 unit (Loupy A et al, BMJ 2019). The software also provides an application for patients allowing secure data transfer (biological analyses, blood pressure, weight). This allows the assessment of the need for additional patient evaluation based on usual monitoring parameters (creatinine, proteinuria) that can be done in the analysis laboratory near the patient's home.

A first evaluation of the use and acceptability among care professionals has been conducted between April and June 2020 and showed excellent results. It is now necessary to obtain real-life data to evaluate the use of the tool among patients and healthcare professionals and its impact on the organisation of care.

This is a prospective interventional study with minimal risks and constraints on the active file of transplant patients followed in ambulatory care for a period of 12 months.

The objective of this study will be to evaluate the use of the Predigraft platform by kidney transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient who received a kidney transplant from a living or a deceased donor and transplanted at least 1 month ago
* Patient over 18 years of age at the time of inclusion
* Stable renal function (glomerular filtration rate>60 mL/min or decision at physician's discretion) at the time of inclusion
* Informed patient with signed consent
* Patient with access to an internet connection with a valid email
* Enrolled in a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Combined transplant (e.g. kidney-heart transplant, kidney-liver transplant)
* Kidney transplant less than 1 month old
* Lack of recovery of kidney function following renal transplantation
* Patient unable to use the telemedicine tool
* Vulnerable participants (minors, protected adults, prisoners)
* Patient under State Medical Assistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-05-25 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who have logged on to the Predigraft application at least 3 times | at 12 months from study inclusion

SECONDARY OUTCOMES:
French version of Functional, Communicative and Critical Health Literacy (FCCHL) scale | at inclusion
  For each subscale of the FCCHL, the literacy score can range from 1 (low) to 5 (high). An overall score is calculated from the scores of the three subscales. A score ≤ 4 corresponds to a low level of literacy.
French version of Functional, Communicative and Critical Health Literacy (FCCHL) | at 12 months after inclusion
  For each subscale of the FCCHL, the literacy score can range from 1 (low) to 5 (high). An overall score is calculated from the scores of the three subscales. A score ≤ 4 corresponds to a low level of literacy.
Connection time | at 12 months after inclusion
Connection frequency | at 12 months after inclusion
Time between two connections | at 12 months after inclusion
Proportion of fonction used | at 12 months after inclusion
Quality of life evaluating using SF36 | at inclusion
  Quality of life evaluated using MOS SF36 questionnaire (Medical Outcomes Study - 36-Item Short Form Health Survey). SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. The SF-36 assesses different dimensions of feeling healthy and well being using 11 questions.These measures rely upon patient self-reporting.. In two dimensions, the answer is binary (yes / no) and in the other 6 in ordinal quality (3 to 6 possible answers). A high score means a better quality of life.
Quality of life evaluating using SF36 | at 6 weeks
  Quality of life evaluated using MOS SF36 questionnaire (Medical Outcomes Study - 36-Item Short Form Health Survey). SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. The SF-36 assesses different dimensions of feeling healthy and well being using 11 questions.These measures rely upon patient self-reporting.. In two dimensions, the answer is binary (yes / no) and in the other 6 in ordinal quality (3 to 6 possible answers). A high score means a better quality of life.
Quality of life evaluated using SF36 | at 12 months
  Quality of life evaluated using MOS SF36 questionnaire (Medical Outcomes Study - 36-Item Short Form Health Survey). SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. The SF-36 assesses different dimensions of feeling healthy and well being using 11 questions.These measures rely upon patient self-reporting.. In two dimensions, the answer is binary (yes / no) and in the other 6 in ordinal quality (3 to 6 possible answers). A high score means a better quality of life.
Medication adherence | at inclusion
  Medication adherence will be evaluation using the Basel Assessment of Adherence Scale Immunosuppression Scale (BAASIS scale). This is a self-assessment scale to evaluate medication adherence.
Medication adherence | at 6 weeks
  Medication adherence will be evaluation using the Basel Assessment of Adherence Scale Immunosuppression Scale (BAASIS scale). This is a self-assessment scale to evaluate medication adherence.
Medication adherence | at 12 months
  Medication adherence will be evaluation using the Basel Assessment of Adherence Scale Immunosuppression Scale (BAASIS scale). This is a self-assessment scale to evaluate medication adherence.
Proportion of hospitalisations | at 12 months after inclusion
Proportion of consultations | at 12 months after inclusion
Proportion of emergency consultations or hospitalisations | at 12 months after inclusion
Overall survival | at 12 months after inclusion
Rejection and dialysis free survival | at 12 months after inclusion
Cumulative incidence of graft rejection | at 12 months after inclusion
Proportion of patients with deteriorated renal function | at 12 months after inclusion
  Renal function deterioration will be defined as an estimated glomerular filtration rate < 30 ml/min/1.73m2 according to the MDRD equation and/or, a 10% decrease between inclusion and 12 months after inclusion.
Probability of graft survival | at inclusion
Probability of graft survival | up to 12 months
Probability of graft survival | at 12 months
Time from date of graft to date of non-protocol DSA | up to 12 months post-inclusion
Time from date of graft to date of non-protocol biopsy | up to 12 months post-inclusion

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital Necker - APHP, Paris
  - Hopital Saint Louis - APHP, Paris

IPD SHARING:
Plan to Share IPD: Undecided